CLINICAL TRIAL: NCT05746871
Title: Post-market Study to Demonstrate the Safety and Performance of an Extension Assist Knee Ankle Foot Orthosis (Agilik) to Improve Gait in Children with Cerebral Palsy
Brief Title: Safety and Performance of Agilik in CP
Acronym: Agilik
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Collaborators: Ro+Ten srl (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: GIP1030
Record Dates: First submitted 2023-02-07; First posted 2023-02-28 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GroupA_Agilik first (Experimental): This arm will be assessed at T0, then it will receive the intervention with Agilik (10 training sessions in 5 weeks) and will perform T1 evaluations, and then it will repeat the evaluations after other 5 weeks (T2) during which they performed they standard care
  Interventions: Device: Agilik; Other: standard care
- GroupB_standard care first (Experimental): This arm will be assessed at T0, then it will continue with their standard care and will perform T1 evaluation after 5 weeks, and then it will receive the intervention with Agilik (10 training sessions in 5 weeks) and the final evaluation (T2)
  Interventions: Device: Agilik; Other: standard care

INTERVENTIONS:
Device: Agilik — The Agilik is a powered orthosis system that can assist or resist motion independently in each gait phase. It is used as a pair of knee-ankle-foot orthosis (KAFO), one for each leg. The device applies up to 12 Nm across the knee in the direction of either flexion or extension. The system consists of an orthosis for each leg integrated with an electro-mechanical actuator, a battery, a carry pack, cabling and application software running on a computer. A foot pressure sensor is embedded in the footbed of the KAFO and connected to the actuator. The foot sensor and angular velocity are used to detect the gait phase of the patient and communicate with the motor controller to provide a unique torque for each gait phase. The torque ramp and intensity can be modified through the Agilik App to cater towards individual patients by assisting or resisting motion during their gait. This allows for the clinician working with the patient to adjust the settings of the device for the patient's needs.
Other: standard care — Subjects will continue with their standard care for 5 weeks

SUMMARY:
The purpose of this post market study is to demonstrate the safety and performance of a powered extension assist (EA) knee ankle foot orthosis (KAFO), or EA-KAFO, in individuals with knee extension deficiency due to cerebral palsy (CP). The EA-KAFO tested in this investigation, whose commercial name is Agilik™, is registered as a Class 1 medical device in the European (EU) Medical Device Regulation (MDR) and with the United States (US) Food and Drugs Administration (FDA). The study will take place in Astrolab at the Istituto Scientifico E. MEDEA - La Nostra Famiglia (IRCCS Medea hereafter). The duration of the investigation will be 36 months. The duration of the study for a single subject will be approximately 10 weeks.

The primary purpose of this study is to demonstrate the safety and performance of a powered extension assist knee ankle foot orthosis (Agilik) in individuals with knee extension deficiency due to cerebral palsy. The focus is on the improvement of anti-gravity knee extension during stance in patients with CP with crouch gait. Therefore, the primary aim is to compare the knee and range of motion (ROM) at baseline and after 10 sessions of Agilik training while wearing Agilik itself. Secondary aim is to compare knee ROM before and after the training with Agilik without wearing Agilik.

The changes in lower extremity functions, kinematics and muscle activity during walking with Agilik compared to baseline conditions will be examined. Furthermore, the performance of Agilik during uphill and downhill walking over the GRAIL platform will be investigated.

Hypotheses when using Agilik:

* Improve knee extension during stance and swing gait phases
* Increase step length, walking distance and speed

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form.
* Stated willingness to comply with all study procedures and availability for the duration of the study, or alternatively, ability to do so based on parent report and physician observation during history and physical examination.
* Age between 5 and 17
* Maximum weight of 70 Kg
* Volunteer who have a gait pathology involving the knee joint, from a diagnosis of CP
* Knee flexion retraction assessed in supine position by less than 10°. Hamstring contracture as assessed by straight leg raising test does not limit ability to participate in the study.
* Subjects must not have had a tibio-tarsal arthrodesis. In addition, they must have at least 10° of passive dorsi-flexion of the ankle.
* Able to walk at least 3 m without stopping with or without a walking aid.
* Able to understand and follow simple directions based on parent report and physician observation during history and physical examination.
* GMFCS level I, II and III
* MAS score ≤ 2

Exclusion Criteria:

* Any neurological, musculoskeletal or cardiorespiratory injury, health condition, or diagnosis other than cerebral palsy that would affect the ability to walk as directed for short periods of time.
* A history of uncontrolled seizure in the past year
* Severe spasticity

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
change of range of motion of the knee overground | 6 weeks
  the range of motion of the knee will be measured by means of BTS Bioengineering S.p.A. optoelectronic system during the overground gait analysis assessment with Agilik
change of range of motion of the knee uphill/downhill | 6 weeks
  the range of motion of the knee will be measured by means of the GRAILoptoelectronic system that is equipped with a motion platform and that will simulate uphill and downhill walking while performing gait analysis assessment with Agilik
change in endurance | 6 weeks
  The endurance will be measured by means of the 6 minute walking test (6MWT) with Agilik
change in gait speed | 6 weeks
  the gait speed will be measured by means of the 10 meters walking test (10mWT) with Agilik
change in spasticity | 6 weeks
  The level of spasticity in the lower limbs will be measured by means of the Ashworth scale (MAS level, Modified Ashworth scale level) with Agilik
change in muscle lengths | 6 weeks
  Joint and muscle lengths examination will be performed manually
change in centre of pressure oscillations | 6 weeks
  Centre of pressure (COP) oscillations will be assessed by means of the force plates embedded in the GRAIL system, during 1 minute of still standing
change in centre of mass oscillations | 6 weeks
  Centre of mass (COM) oscillations will be measured during 1 minute of standing by means of the G-Sensor, a wearable three axial accelerometer and gyroscope
satisfaction using Agilik | 6 weeks
  the children's satisfaction with Agilik will be evaluated with the Quebec User Evaluation of Satisfaction adapted to children (QUEST 2.1).

SECONDARY OUTCOMES:
change of range of motion of the knee overground without Agilik | 6 weeks
  the range of motion of the knee will be measured by means of BTS Bioengineering S.p.A. optoelectronic system during the overground gait analysis assessment without Agilik
change of range of motion of the knee uphill/downhill without Agilik | 6 weeks
  the range of motion of the knee will be measured by means of the GRAILoptoelectronic system that is equipped with a motion platform and that will simulate uphill and downhill walking while performing gait analysis assessment without Agilik
change in endurance without Agilik | 6 weeks
  The endurance will be measured by means of the 6 minute walking test (6MWT) without Agilik
change in gait speed without Agilik | 6 weeks
  the gait speed will be measured by means of the 10 meters walking test (10mWT) without Agilik
change in centre of pressure oscillations without Agilik | 6 weeks
  Centre of pressure (COP) oscillations will be assessed by means of the force plates embedded in the GRAIL system, during 1 minute of still standing without Agilik
change in centre of mass oscillations without Agilik | 6 weeks
  Centre of mass (COM) oscillations will be measured during 1 minute of standing without Agilik by means of the G-Sensor, a wearable three axial accelerometer and gyroscope

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Medea, Bosisio Parini, Italy

IPD SHARING:
Plan to Share IPD: No